CLINICAL TRIAL: NCT05666947
Title: Effectiveness of Two Exercises in Preventing Lower-Limb Lymphedema After Gynecological Cancer Surgery: a Randomized Controlled Trial
Brief Title: Effectiveness of Two Exercises in Preventing Lower-Limb Lymphedema After Gynecological Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Yun Hsu (Other)
Responsible Party: Sponsor-Investigator, Yu-Yun Hsu, Professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-ER-105-444
Record Dates: First submitted 2022-12-02; First posted 2022-12-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2022-12

CONDITIONS: Lymphedema of Leg; Gynecologic Cancer; Exercise
Keywords: Elastic-band; Gynecological cancer; Lymphedema; Quality of life; Resistance exercise; Self-management
MeSH Terms: conditions — Motor Activity; Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based resistance exercise (Experimental): The experimental group participated in a home-based exercise program for eight weeks, namely elastic-band resistance exercise. Participants were forwarded to the next exercise session every two weeks and completed the exercise program within eight weeks. The program included upper and lower limb exercises. The home-based exercise program contained four sessions, namely: warm-up, start-up, vigorous, and reinforcement sessions. Participants received guidelines from a booklet and video about elastic-band resistance.
  Interventions: Other: Home-based exercise
- Non-resistance exercise (Placebo Comparator): The control group participated in an exercise program for eight weeks, namely conventional non-resistance exercise, which contained four sessions: warm-up, start-up, vigorous, and reinforcement. Participants were forwarded to the next exercise session every two weeks and completed the exercise program within eight weeks. Participants in the control group received guidelines from a booklet and video about the conventional non-resistance exercise.
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Home-based exercise — Eight weeks of home-based exercise programs

SUMMARY:
Background:

Lower-limb lymphedema is one of the complications after gynecological cancer surgery. Patients with lymphedema are more likely to limit their daily life activities and become inactive, leading to negative influences on quality of life. Although studies on resistance exercise primarily focus on the upper limb, there scarce evidence of the application of this exercise to the lower limb has been reported.

Objective:

This study will aim to compare the effect of resistance and non-resistance exercises in the prevention of lower-limb lymphedema, increasing self-management, and improving the quality of life of the patients following gynecological cancer surgery.

Design:

A single-blinded randomized controlled trial.

Settings and participants:

Sixty patients with gynecological cancer will recruit from a gynecological ward and will be randomly assigned to the elastic-band resistance exercise group (experimental group, n = 30) or conventional non-resistance exercise group (control group, n = 30).

Methods:

Both groups will receive one-to-one training about upper and lower limb exercises within 1 week after surgery. Each exercise will consist of a 5-minute warm-up session, a 20-minute main session, and a relaxing session. Patients in the experimental group will use an elastic band and change the elastic band from low to medium resistance. Patients in the experimental and control groups will receive guidelines from a booklet and video about elastic-band resistance and conventional non-resistance exercise, respectively. All patients will be evaluated at three-time points: T0-within 1 week after surgery and before the intervention, T1-10-11 weeks after surgery and within 1 week after intervention, T2-3 months after intervention using Lymph-ICF-LL scale, EORTC QLQ-C30 questionnaire, limb circumference measurements, and lymph self-management questionnaire. The Chi-square test, Fisher's exact test, the Mann-Whitney U-test, and the Generalized Estimating Equations will be used for the statistical analysis of the data.

Anticipated Outcomes: Findings from this study could provide a reference for home-based resistance exercise guidelines and be integrated into the care of activities for women following gynecological surgery with lower-limb lymphoedema.

DETAILED DESCRIPTION:
1. Participants and setting Participants were recruited from a gynecological ward of a medical center in southern Taiwan. The following criteria were used to determine who was eligible to participate in this study: (1) women who planned to undergo gynecological cancer surgery with lymphadenectomy, and (2) at least 20 years old. Exclusion criteria for the participants were: (1) heart failure; (2) renal failure; (3) cardiovascular accident; (4) abscess or infection in legs; or (5) psychological disorders.
2. Sample size G-power software version 3.1.9 was applied to estimate the sample size. The sample size was determined based on a previous study. Given an α-level of 0.05, an effect size of 0.37, a power of 0.80, and considering a 15% possibility of participants' dropping out, the minimum required sample size was estimated as 30 participants in each group.
3. Randomization and Blinding Eligible participants were randomly assigned into either an experimental group or a control group using a randomized block design with a ratio of 2:2. A research staff who was not involved in data collection generated in advance the random allocation sequence with 15 blocks. Each block contributed to the allocation of 2 participants in the experimental group (anti-resistance exercise) and 2 participants in the intervention group. Sequential numbers which assigned to two groups were generated and placed in sealed opaque envelopes.
4. Data analysis Data were managed and analyzed using SPSS. Descriptive statistics were applied to summarize the characteristics of the participants and study outcomes. Chi-square tests (or Fisher's exact test) and Mann-Whitney U-test were applied for the group comparisons in demographic data and outcome variables and at baseline. The Generalized Estimating Equations (GEE) were used to assess for any differential changes in the outcome variables by testing the time effect, group effect, and group*time effect with p < 0.05 as a level of significance.
5. Ethical considerations Before data collection, the hospital's Institutional Review Board of the primary investigator reviewed and approved this study (IRB No. B-ER-105-444).

ELIGIBILITY:
Inclusion Criteria:

* women who planned to undergo gynecological cancer surgery with lymphadenectomy
* at least 20 years old

Exclusion Criteria:

* heart failure
* renal failure
* cardiovascular accident
* abscess or infection in legs
* psychological disorders

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
lymphoedema-related quality of life | Three-time points, (1) baseline(T0), (2) change from baseline at 2 months(T1), (3) change from baseline at 5 months(T2).
  Chinese version of the Lymph-ICF-LL(Lymphoedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphoedema) was used to evaluate the quality of life related to lower-limb lymphedema. This scale includes 28 questions over five domains: physical function (6 questions), mental function (6 questions), general tasks/household (3 questions), mobility (7 questions), and life/ social life (6 questions). The participants were required to rate their answers on an 11-point scale (from 0 = no problem to 10 = very serious). The total score and scores on each domain of the Lymph-ICF-LL were computed as follows: (sum of scores on questions/ total number of answered questions) x 10. Thus, the scores ranged from 0 to 100 with a higher score indicating lower quality of life related to lower limb lymphedema.
cancer quality of life | Three-time points, (1) baseline(T0), (2) change from baseline at 2 months(T1), (3) change from baseline at 5 months(T2).
  The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3 was used to measure the quality of life related to cancer. The questionnaire contained 30 questions, including five functional items (physical, role, emotional, cognitive, and social functioning), nine symptom items, and the single item of global health status. Except for the global health status, each question was rated from 1 (not at all) to 4 (very much). In addition, the global health status was rated from 1 (very poor) to 7 (excellent).
limb circumference measurement | Three-time points, (1) baseline(T0), (2) change from baseline at 2 months(T1), (3) change from baseline at 5 months(T2).
  The bilateral circumferences of lower extremities were measured to assess the lymphedema status.

SECONDARY OUTCOMES:
Lymph self-management | Three-time points, (1) baseline(T0), (2) change from baseline at 2 months(T1), (3) change from baseline at 5 months(T2).
  The Lymph Self-management Scale, developed by the authors, was used to measure the participants' self-management of lymphedema in the past two weeks. The self-reported questionnaire contained 20 questions including self-examination for limb edema, wearing comfortable shoes, eating protein-rich foods, avoiding spicy or caffeinated foods, keeping regular exercise, avoiding long-time standing or sitting (> 1 hour), skin protect, and weight control. Each question was scored from 1 (never) to 5 (always). Scores range from 20 to 100, a higher score indicating better lymph self-management.
Exercise adherence | at T1 (10-11 weeks after surgery and within 1 week after intervention completion)
  A dialog about exercise frequency weekly and total exercise time weekly was designed to measure the exercise adherence of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Yun Hsu, Principal Investigator — National Cheng Kung University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu YY, Lin CF, Liang PC, Nguyen TTB, Hsu KF. Effects of resistance exercise on reducing the risk of lower-limb lymphedema after gynecological cancer surgery. Asia Pac J Oncol Nurs. 2025 Jul 14;12:100756. doi: 10.1016/j.apjon.2025.100756. eCollection 2025 Dec. PMID 40821966